CLINICAL TRIAL: NCT02584699
Title: Phase II Study of Stereotactic Ablative Radiotherapy in Elderly Patients With Stage I Non-Small Cell Lung Cancer
Brief Title: Study of Stereotactic Ablative Radiotherapy (SABR) in Elderly Stage I NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luhua Wang (Unknown)
Responsible Party: Sponsor-Investigator, Luhua Wang, Deputy president, Cancer Hospital, Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33320140105
Record Dates: First submitted 2015-08-13; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SABR (Experimental): SABR group includes patients receiving pre-identified fractionated Stereotactic Ablative Radiotherapy (SABR)
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — Six Gy irradiation per fraction times 12 fractionations, resulting a total dose of 72Gy
  Other Names: Stereotactic body radiation therapy (SBRT)

SUMMARY:
This study aims to prospectively investigate the efficacy, toxicity and quality of life (QOF) of stereotactic ablative radiotherapy (SABR) using a moderate fractionation of 72 Gy/6 Gy/12 F (BED10 = 115 Gy) in a single arm of elderly ( ≥ 70) patients with stage I (2009 UICC) non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This study aims to prospectively investigate the local regional control, overall survival, treatment related toxicities and quality of life (QOF) of elderly stage I NSCLC patients receiving stereotactic ablative radiotherapy (SABR) with a moderate fractionation of 72 Gy/6 Gy/12 F (BED10 = 115 Gy). Patients' general characteristics, treatment modality, dose-volume histogram (DVH) parameters, toxicity profiling, quality of life, pattern of failure as well as survival time will be prospective recorded for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70
* Pathologically or cytologically confirmed NSCLC
* Stage T1- 2 N0M0 based on adequate workup
* Peripheral tumor
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Inoperable NSCLC

Exclusion Criteria:

* Pathologically or cytologically confirmed SCLC
* Direct evidence of regional or distant metastasis
* Central tumor
* Past history of malignancy
* Past history of thoracic irradiation
* Past history of chemotherapy
* Past history of thoracic surgery
* Pure Bronchioalveolar adenocarcinoma
* Active systemic, pulmonary or pleural lung diseases
* Pulmonary infection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Local regional progression free survival | 2 year
  Duration between radiotherapy commencement and local progression, regional progression, death of cancer or last date of follow up.

SECONDARY OUTCOMES:
Objective response rate | 1 month after RT
  Tumor response to radiotherapy evaluated by RECIST 1.1
Progression free survival | 2 year
  Duration between radiotherapy commencement and any progression, death of cancer or last date of follow up.
Overall survival | 2 year
  Duration between radiotherapy commencement and any cause of death or last date of follow up.
Grade ≥ 2 radiation induced normal tissue toxicity | 1 year
  Incidence of radiation induced toxicities on lung, oesophagus, rib or chest wall pain assessed by CTCAE v 4.0
Questionnaire on quality of life | 2 year
  Physical and psychologic status assessed by specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jingbo Wang, Dr., Principal Investigator — Cancer Hospital/Institute, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital/Institute, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Havlik RJ, Yancik R, Long S, Ries L, Edwards B. The National Institute on Aging and the National Cancer Institute SEER collaborative study on comorbidity and early diagnosis of cancer in the elderly. Cancer. 1994 Oct 1;74(7 Suppl):2101-6. doi: 10.1002/1097-0142(19941001)74:7+3.0.co;2-m. PMID 8087777
- [Background] Yang L, Li L, Chen Y, Parkin DM. [Mortality time trends and the incidence and mortality estimation and projection for lung cancer in China]. Zhongguo Fei Ai Za Zhi. 2005 Aug 20;8(4):274-8. doi: 10.3779/j.issn.1009-3419.2005.04.05. Chinese. PMID 21108881
- [Background] Wingo PA, Cardinez CJ, Landis SH, Greenlee RT, Ries LA, Anderson RN, Thun MJ. Long-term trends in cancer mortality in the United States, 1930-1998. Cancer. 2003 Jun 15;97(12 Suppl):3133-275. doi: 10.1002/cncr.11380. PMID 12784323
- [Background] Raz DJ, Zell JA, Ou SH, Gandara DR, Anton-Culver H, Jablons DM. Natural history of stage I non-small cell lung cancer: implications for early detection. Chest. 2007 Jul;132(1):193-9. doi: 10.1378/chest.06-3096. Epub 2007 May 15. PMID 17505036
- [Background] Rowell NP, Williams CJ. Radical radiotherapy for stage I/II non-small cell lung cancer in patients not sufficiently fit for or declining surgery (medically inoperable): a systematic review. Thorax. 2001 Aug;56(8):628-38. doi: 10.1136/thorax.56.8.628. PMID 11462066
- [Background] Dosoretz DE, Galmarini D, Rubenstein JH, Katin MJ, Blitzer PH, Salenius SA, Dosani RA, Rashid M, Mestas G, Hannan SE, et al. Local control in medically inoperable lung cancer: an analysis of its importance in outcome and factors determining the probability of tumor eradication. Int J Radiat Oncol Biol Phys. 1993 Oct 20;27(3):507-16. doi: 10.1016/0360-3016(93)90373-4. PMID 8226142
- [Background] Timmerman R, Paulus R, Galvin J, Michalski J, Straube W, Bradley J, Fakiris A, Bezjak A, Videtic G, Johnstone D, Fowler J, Gore E, Choy H. Stereotactic body radiation therapy for inoperable early stage lung cancer. JAMA. 2010 Mar 17;303(11):1070-6. doi: 10.1001/jama.2010.261. PMID 20233825
- [Background] Senthi S, Lagerwaard FJ, Haasbeek CJ, Slotman BJ, Senan S. Patterns of disease recurrence after stereotactic ablative radiotherapy for early stage non-small-cell lung cancer: a retrospective analysis. Lancet Oncol. 2012 Aug;13(8):802-9. doi: 10.1016/S1470-2045(12)70242-5. Epub 2012 Jun 22. PMID 22727222